CLINICAL TRIAL: NCT07065123
Title: Study on Atrioventricular and Bundle Branch Block Vulnerability Identified by Outcome-based Risk Modeling （the SAVIOR Study）
Brief Title: Study on Heart Block Risks Using Outcome-Based Modeling
Acronym: SAVIOR
Status: Completed | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jingfeng Wang, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: AS-TAVR-2023-04-10
Record Dates: First submitted 2025-06-26; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Left Bundle-Branch Block; Aortic Stenosis
Keywords: Transcatheter Aortic Valve Replacement; Permanent Pacemaker Implantation; Left Bundle Branch Block; Predictive Model
MeSH Terms: conditions — Bundle-Branch Block; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Permanent pacemaker implantation after TAVR surgery
  Interventions: Other: The population undergoing TAVR for aortic valve stenosis with outcomes of permanent pacemaker implantation and complete left bundle branch block after surgery
- Complete left bundle branch block occurred after TAVR surgery
  Interventions: Other: The population undergoing TAVR for aortic valve stenosis with outcomes of permanent pacemaker implantation and complete left bundle branch block after surgery

INTERVENTIONS:
Other: The population undergoing TAVR for aortic valve stenosis with outcomes of permanent pacemaker implantation and complete left bundle branch block after surgery — The population undergoing TAVR for aortic valve stenosis with outcomes of permanent pacemaker implantation and complete left bundle branch block after surgery

SUMMARY:
This study developed a prediction model for high-grade atrioventricular block (AVB) and complete left bundle branch block (CLBBB) following transcatheter aortic valve replacement (TAVR) in Chinese patients with aortic stenosis (AS). Analyzing 112 patients from Sun Yat-sen Memorial Hospital (2017-2024), the study incorporated clinical, electrocardiographic, and procedural variables to identify risk factors via logistic regression. A nomogram was constructed and validated internally (bootstrapping) and externally (temporal validation), with performance assessed using AUC, C-index, and calibration tests. The model aims to improve preoperative risk stratification and guide individualized management for TAVR-related conduction disturbances in this understudied population. Analyses were conducted in R 4.2.3 (significance: *p* < 0.05).

DETAILED DESCRIPTION:
In recent years, transcatheter aortic valve replacement (TAVR) has emerged as a minimally invasive surgical approach and has gradually become a standard treatment option for patients with moderate to severe aortic stenosis（AS), particularly those at high surgical risk or deemed ineligible for conventional surgery. TAVR has been widely adopted in clinical practice.

However, post-TAVR cardiac conduction disturbances are among the most frequently observed complications, particularly complete left bundle branch block (CLBBB) and high-degree atrioventricular block (AVB) requiring permanent pacemaker implantation (PPI). These complications are associated with an increased risk of heart failure and cardiac mortality. Identified risk factors include patient-specific characteristics, electrocardiographic features, intraoperative procedural techniques, and the type of device used.

Current research on post-TAVR conduction disorders predominantly focuses on Western populations. However, Chinese AS patients exhibit distinct clinical features-such as higher degrees of valve calcification and a higher prevalence of bicuspid aortic valves-which may lead to differences in risk factors for conduction abnormalities. Moreover, prior studies have largely focused on isolated risk factors rather than developing integrated models to quantify the risk of such complications. Against this backdrop, the purpose of this study is to address the knowledge gap in postoperative risk prediction for Chinese patients. By constructing a risk prediction model tailored to Chinese AS patients for post-TAVR cardiac conduction block, we aim to improve preoperative risk assessment and individualized clinical management, thereby providing actionable guidance for clinical decision-making.

This study included 112 aortic stenosis patients undergoing TAVR at Sun Yat-sen Memorial Hospital (2017-2024), divided into internal (2017-2022) and external (2023-2024) validation cohorts.

Data covered demographics, medical history, ECG, echocardiography, biomarkers, and valve parameters. Outcomes were permanent pacemaker implantation (PPI) ≤48h post-TAVR and complete left bundle branch block (CLBBB).

Univariate logistic regression (p<0.20 threshold) and stepwise multivariate analysis (R "MASS" package, AIC-based) identified predictors for nomogram development. Model performance was assessed via AUC, C-index, ROC, and Hosmer-Lemeshow test. Internal validation used 1000 bootstrap resamples; external validation employed temporal validation. Analyses were performed in R 4.2.3 (significance: p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) with severe symptomatic aortic stenosis (AS) meeting 2021 ESC/EACTS Guidelines and Chinese Expert Consensus criteria (AVA <1.0 cm², or peak jet velocity ≥4.0 m/s, or mean gradient ≥40 mmHg)
* Scheduled to undergo transcatheter aortic valve replacement (TAVR) in Sun Yat-Sen Memorial Hospital

Exclusion Criteria:

* Pre-existing complete left bundle branch block (CLBBB) on baseline ECG
* Patients with pre-existing permanent pacemaker implantation
* Inability to comply with follow-up protocol

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This single-center retrospective study enrolled 112 consecutive patients with aortic stenosis (AS) who underwent TAVR at the Department of Cardiology, Sun Yat-sen Memorial Hospital between January 2017 and December 2024. The cohort was divided into:
  Internal validation cohort: Patients treated from 2017 to 2022 (n=68)
  External validation cohort: Patients treated from 2023 to 2024 (n=44)
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Permanent Pacemaker Implantation Rate for High-Grade AVB (≥Mobitz II/3°) Post-TAVR (12-Lead ECG Confirmed) | 7 years
  Number of participants requiring permanent pacemaker implantation (PPI) due to high-grade atrioventricular block (AVB; ≥2nd degree Mobitz II or 3rd degree) within 48 hours post-TAVR, as clinically indicated and confirmed by 12-lead ECG and cardiology consultation
Complete left bundle branch block rate post-TAVR (12-lead ECG confirmed) | 7 years
  Number of participants developing new complete left bundle branch block , as defined by standard ECG criteria (QRS duration ≥120ms with characteristic morphology), within 48 hours post-transcatheter aortic valve replacement.

IPD SHARING:
Plan to Share IPD: No